CLINICAL TRIAL: NCT02379364
Title: Effectiveness of Diacutaneous Fibrolysis Technique on Pain, Range of Motion, Strength and Function in Patients With Patellofemoral Pain Syndrome
Brief Title: Diacutaneous Fibrolysis and Patellofemoral Pain Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Pablo Fanlo Mazas, Unidad de Investigación en Fisioterapia, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI/01
Record Dates: First submitted 2015-02-09; First posted 2015-03-04 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Physiotherapy; Patellofemoral Pain Syndrome; Manual therapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): Diacutaneous Fibrolysis treatment
  Interventions: Device: Diacutaneous Fibrolysis

INTERVENTIONS:
Device: Diacutaneous Fibrolysis — Diacutaneous Fibrolysis is a non invasive physiotherapeutic technique applied by means a set of metallic hooks having the advantage of allowing a deeper and more precise application, which could not be achieved manually

SUMMARY:
The aim of the study will be to assess the effectiveness of Diacutaneous Fibrolysis technique on pain, range of motion (Patellofemoral joint mobility test and muscle length test), strength and function in patients with Patellofemoral Pain Syndrome and muscle shortening.

Muscle imbalance is one of most important factor associated with Patellofemoral Pain Syndrome. Shortening of lateral muscles of the thigh have a close relationship with patella position and tracking and patellofemoral pain. The scientific evidence for effectiveness of any soft tissue mobilization technique in patellofemoral pain syndrome patients is poor.

Diacutaneous Fibrolysis is a non-invasive physiotherapeutic technique to release adherences and fibrosis between the different musculoskeletal structures. Diacutaneous Fibrolysis is applied by a set of metallic hooks having the advantage of allowing a deeper and more precise application, which could not be achieved manually.

The present study evaluates the effectiveness of Diacutaneous Fibrolysis technique applied in the soft tissues more related with patellofemoral pain.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral patellofemoral pain longer than three months
* Anterior or retropatellar pain of non-traumatic origin that is provoked by at least two of the following activities: prolonged sitting or kneeling, squatting, running, hopping, jumping, or stair ascending/descending.
* The presence of pain on palpation of the patellar facets, on step down from 25 cm step, or during a double leg squat.
* Pain over the previous week equal to or greater than 3 on a 10-cm visual analogue scale.
* The presence of muscle shortening in rectus femoris or tensor fascia lata muscle length test and/or hypo-mobility or stiffness in the compartmental muscle play.

Exclusion Criteria:

* Previous knee surgery or traumatic lesions
* Concomitant injury or pathology of other knee structures
* History of patella subluxation or dislocation
* Evidence of knee joint effusion
* Pain in and/or referred from the hip or lumbar spine
* Currently undergoing physiotherapy treatment for Patellofemoral pain syndrome or use anti-inflammatories or corticosteroid medication at the same time of the study.
* Subjects unable or unwilling to give informed to written consent or fulfil questionnaires.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain intensity | 2 weeks
  Visual analogue scale (VAS)

SECONDARY OUTCOMES:
Pressure Pain Threshold | 2 weeks
  Pressure algometry
Muscle Length Test | 2 weeks
  Range of motion measured by digital inclinometer in hip adduction for iliotibial band, knee flexion for rectus femoris muscle and knee extension for hamstrings muscles
Isometric Strength of Quadriceps Muscle | 2 weeks
  digital dynamometer
Functional Capacity | 2 weeks
  Unilateral squat test and step test for assessing functional capacity
Functional Status and disability | 2 weeks
  Anterior Knee Pain Scale
Global Rating of Change Scale | 2 weeks
  global improvement on a five point Likert scale and visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Fanlo, PhD, Principal Investigator — Unidad de Investigación en Fisioterapia. Universidad de Zaragoza
Locations (1):
- Unidad de Investigación en Fisioterapia. Universidad de Zaragoza, Zaragoza, Spain